CLINICAL TRIAL: NCT01251822
Title: Double-dummy, Double-blind, Randomised, Parallel Group, Controlled Comparative Study of Polyethylene Glycol (PEG)Plus Electrolytes Versus Prucalopride in Females With Chronic Constipation Who Failed Adequate Relief With Laxatives
Brief Title: Comparator Study of PEG 3350 Versus Prucalopride in Females With Chronic Constipation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Norgine (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PEG-01/2010 (PRUC)
Record Dates: First submitted 2010-11-30; First posted 2010-12-02 (Estimated); Last update posted 2012-08-31 (Estimated); Status verified 2012-08

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation | interventions — polyethylene glycol 3350; Electrolytes; prucalopride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PEG 3350 (Experimental): PEG 3350 plus electrolytes in solution plus placebo tablets
  Interventions: Drug: PEG 3350 plus electrolytes
- Prucalopride (Active Comparator): Prucalopride tablets plus placebo solution
  Interventions: Drug: Prucalopride

INTERVENTIONS:
Drug: PEG 3350 plus electrolytes — Each sachet of PEG 3350 is dissolved in 125 mL of water. Patients receive two sachets of PEG 3350 plus electrolytes followed by two placebo tablets for the first 14 days, after which dosage adjustment is permitted, according to effect. Each patient is treated for 28 days in total.
  Arms: PEG 3350
Drug: Prucalopride — Patients less than 65 years of age receive a solution containing two sachets of reconstituted placebo followed by two prucalopride 1 mg tablets for 28 days.
  Patients more than 65 years of age receive a solution containing two sachets of reconstituted placebo followed by one prucalopride 1 mg tablet and one placebo tablet for 28 days.
  Arms: Prucalopride

SUMMARY:
This study is to compare the efficacy and safety of polyethylene glycol (PEG) 3350 with that of prucalopride in the treatment of chronic constipation in females. A total of 240 patients will be randomly allocated to treatment with one or the other agent. The study consists of a 14-day run-in period, with treatment subsequently administered for 28 days on a daily basis. During the study, patients will fill in a stool diary, samples of faeces will be collected, and colonic transit time will be measured prior to therapy, and from days 22 to 28 of treatment. The proportion of patients with normalised bowel movements (three or more spontaneous movements) during the last week of the study (days 22 to 28 of treatment) will be compared between treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Patient's written informed consent must be obtained prior to inclusion.
2. Female patient aged 18 to 75 years with chronic constipation confirmed during the run-in period.
3. Patient with a history of self-reported chronic constipation for at least 6 months and not satisfied with laxatives in the past. Chronic constipation is defined by ROME III criteria (Drossman DA et al., 2006; Drossman DA, 2006) and characterised by:

   * <3 successful bowel movements per week and at least 1 of the following symptoms that has to have been present for at least 3 months prior to enrolment:

     * Straining in at least 25% of defecations.
     * Lumpy or hard stools in at least 25% of defecations.
     * Sense of incomplete evacuation in at least 25% of defecations.
     * Sensation of anorectal blockage in at least 25% of defecations.
     * Manual manoeuvres to facilitate at least 25% of defecations.
4. Less than 3 SCBMs during the last week of the run-in period.
5. Willing and able to follow the entire procedure and to comply with study instructions.

Exclusion Criteria:

1. History or evidence of organic disease in the large bowel, intestinal perforation or obstruction due to structural or functional disorder of the gut wall, ileus, severe inflammatory conditions of the intestinal tract such as Crohn's disease or ulcerative colitis, toxic megacolon or occlusive or subocclusive syndrome.
2. Abdominal pain of unknown cause.
3. Known allergy to PEG 3350, prucalopride or known hypersensitivity to any of the other study medication ingredients.
4. Drug or alcohol abuse (recent history or within previous 12 months).
5. Pregnant or lactating female.
6. Severe or acute disease within the last 2 weeks prior to the start of the study based on Investigator's judgement.
7. Use of:

   * Any oral purgatives/laxatives and prokinetics within the last 14 days prior to dosing and during the study.
   * Any opioids, anticholinergics, tricyclic anti-depressants, monoamine-oxidase inhibitors or iron preparations within the last 4 weeks prior to dosing.
   * Any calcium-antagonists, beta-blockers or diuretics within the last 4 weeks prior to dosing.
   * Other investigational drugs or prescribed medications affecting gastrointestinal function such as antispasmodics, drugs affecting motility (e.g. erythromycin), anthraquinones, ondansetron or other 5-hydroxytryptamine-3 (5-HT3) antagonists.
   * Any other medication which in the opinion of the investigator could interfere with the principal function of the gastrointestinal tract.
8. Insufficient documentation of chronic constipation during the run-in period.
9. Diarrhoea during the run-in period.
10. Anamnesis/medical history with clinically relevant findings in the gastrointestinal tract during proctoscopy, colonoscopy, sigmoidoscopy or computer tomography, or any other condition which in the Investigator's opinion, may put the patient at significant risk, may confound the study results or may interfere significantly with the results of the study.
11. Participation in another clinical study of drugs or devices parallel to or less than 90 days before study entry or previous participation in this study.
12. Gastrointestinal surgery within the last 6 months prior to the start of the study.
13. Malignant tumours within the last 5 years prior to the start of the study.
14. Uncontrolled blood pressure or terminal cardiac, liver and/or kidney diseases.
15. Patient with diagnosis or evidence of the following diseases: hypothyroidism, diabetes mellitus, porphyria, pituitary gland insufficiency, pheochromocytoma, glucagonoma, neurological diseases (e.g. Hirschprung diseases, neurofibromatosis, Chagas diseases, stroke, autonomous neuropathy, intestinal pseudo-obstruction, multiple sclerosis, medullar injury, Parkinson diseases, Shy-Drager syndrome), collagenosis, vasculitis, myopathy (e.g. sclerodermatitis, amyloidosis, dermatomyositis), intoxication with heavy metals (e.g. lead, phosphorus, arsenic, mercury).
16. Patients with known HIV infection.
17. Woman of childbearing potential, who is not using and not willing to use medically reliable methods of contraception for the entire study duration, such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices, unless she is surgically sterilised/hysterectomised or any other criteria considered sufficiently reliable by the Investigator in individual cases.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2010-11; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Number of spontaneous bowel movements | Days 22 to 28 of treatment
  Proportion of patients having normal number of spontaneous bowel movements during the last treatment week.

CONTACTS AND LOCATIONS:
Overall Officials: Rodica Cinci, Prof Dr, Principal Investigator — Pierrel Research
Locations (1):
- Pierrel Research, Timișoara, Romania

REFERENCES:
- [Derived] Cinca R, Chera D, Gruss HJ, Halphen M. Randomised clinical trial: macrogol/PEG 3350+electrolytes versus prucalopride in the treatment of chronic constipation -- a comparison in a controlled environment. Aliment Pharmacol Ther. 2013 May;37(9):876-86. doi: 10.1111/apt.12278. Epub 2013 Mar 11. PMID 23480216